CLINICAL TRIAL: NCT05748743
Title: Using a Randomized Control Trial to Evaluate the Effectiveness of Glove Changing in Reducing Wound-related Complications Following Cesarean Section in Vietnam
Brief Title: Effectiveness of Glove Changing in Reducing Wound-related Complications
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hung Vuong Hospital (Other)
Responsible Party: Principal Investigator, Tri Bao Nguyen, Principle investigator, Hung Vuong Hospital
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: CK62721303
Record Dates: First submitted 2023-02-18; First posted 2023-03-01 (Actual); Last update posted 2023-03-02 (Actual); Status verified 2023-02

CONDITIONS: Wound Complication
Keywords: Complications; Glove changing; Eesarean surgery; Infections; Vietnam
MeSH Terms: conditions — Infections

STUDY DESIGN:
Intervention Model Description: The study is a parallel-group randomized control trial with 2 arms. Arm 1 includes patients who will have glove changed prior to abdominal closure during cesarean surgery. Aim 2 includes patients who will not have glove changed prior to abdominal closure during cesarean surgery. All patients are randomized using computer-generated sequences with allocation ratio 1:1. Clinic visits are performed at 2 time points. Visit 1 is at 2-3 days post-surgery and visit 2 is at 30 ± 2 days post-surgery where primary and secondary outcomes are measured. The primary outcomes of interest are any wound complications occurring after the surgery, including seroma, hematoma, wound separation, and wound infection. Secondary outcomes are any signs of SSI, including fever, swelling, redness, and pain surrounding the incisional area. The outcomes will be evaluated during clinic visits by qualified medical practitioners who are blind to the intervention group assignment.
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: Participants, investigators, and outcomes assessor are blind to the intervention group assignment.The only people that were unmasked were the surgical team.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Glove change group (Experimental): The surgical gloves were changed prior to closure of the peritoneum or closure of the abdominal fascia
  Interventions: Procedure: glove changing
- Usual care group (No Intervention): The surgical gloves were not changed before abdominal closure

INTERVENTIONS:
Procedure: glove changing — Surgical gloves were changed prior to abdominal closure during Cesarean section to evaluate its effectiveness in reducing wound complications after surgery
  Arms: Glove change group

SUMMARY:
This study aimed to investigate the effectiveness of glove changing in reducing complications of cesarean deliveries in Vietnam.

DETAILED DESCRIPTION:
In Vietnam, the rate of Cesarean section (CS) is very high, ranging from 40-50%. Despite that, there are very limited publications concerning the risk factors, complications, and management of surgical site infection (SSI) following CS. Our study is the first to investigate the effectiveness of glove changing in reducing the incidence of post-operative infections in Vietnam. Specifically, the aims of this study are 1) to evaluate whether changing gloves during CS reduces complications and SSI, and 2) to identify other factors that are associated with complications and SSI.

ELIGIBILITY:
Inclusion criteria

* pregnant women were 18 years old or higher;
* pregnant women had cesarean surgery performed at Hung Vuong hospital;
* pregnant women lived close to Ho Chi Minh city and agreed to return for postpartum care one-month post-surgery.

Exclusion criteria

* pregnant women had fever during labor;
* pregnant women had systemic infectious conditions;
* pregnant women had surgical site infection SSI or sexually infectious conditions;
* pregnant women had ongoing internal conditions such as pre-eclampsia, severe anemia, American Society of Anesthesiologists (ASA) ≥ 3, New York Heart Association (NYHA) class 3 or above, pulmonary edema, or severe asthma.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — We only recruited pregnant women to participate in this study
Enrollment: 678 (Actual)
Dates: Start 2020-12-18 (Actual); Primary Completion 2021-02-25 (Actual); Study Completion 2021-02-25 (Actual)

PRIMARY OUTCOMES:
Wound complications | Within 4 weeks after surgery
  Seroma, hematoma, wound separation, and wound infection

SECONDARY OUTCOMES:
Surgical site infection | Within 4 weeks after surgery
  Fever, swelling, redness, and pain surrounding the incisional area

CONTACTS AND LOCATIONS:
Overall Officials: Tuyet Hoang, Doctor, Study Director — Hung Vuong Hospital
Locations (1):
- Hung Vuong hospital, Ho Chi Minh City, Vietnam

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-09-14): https://cdn.clinicaltrials.gov/large-docs/43/NCT05748743/Prot_SAP_000.pdf